CLINICAL TRIAL: NCT02508415
Title: Relationship Between Obesity and Periodontal Disease
Acronym: ROPD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Malaya (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: UMalaya
Record Dates: First submitted 2015-04-02; First posted 2015-07-27 (Estimated); Last update posted 2015-07-27 (Estimated); Status verified 2015-07

CONDITIONS: Obese; Periodontal Disease
Keywords: obesity; periodontal disease; intervention
MeSH Terms: conditions — Obesity; Periodontal Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Non Surgical Periodontal Therapy (Experimental): Will receive oral hygiene education, scaling and root planing. OHE includes brushing and flossing techniques, chlorhexidine mouth rinse twice a day
  Interventions: Other: Non Surgical Periodontal Therapy
- No Non Surgical Periodontal Therapy (No Intervention): No treatment received

INTERVENTIONS:
Other: Non Surgical Periodontal Therapy — OHE, scaling root planing, mouth wash
  Arms: Non Surgical Periodontal Therapy

SUMMARY:
Obesity is an epidemic with increasing prevalence in the Asia Pacific region. The first Malaysian national estimate in 1996 of obesity was 5.8%. A systematic review reported a marked increase in obesity in 2003, 2004 and 2006 with 12.2%, 12.3% and 14.0% respectively.

Periodontal disease is a chronic inflammatory disease which results in gingival inflammation, irreversible attachment loss, alveolar bone destruction and eventually tooth loss. Worldwide, the prevalence of periodontitis in the adult population is about 10-15%. Periodontal disease, through inflammation and destruction of the periodontium produces clinical signs and symptoms, some of which may have a considerable impact on quality of life (QoL).

A positive association between obesity and periodontal disease was repeatedly demonstrated worldwide. Obese individuals have elevated levels of circulating TNF- α and IL-6 compared to normal weight individuals. These cytokines decrease after weight loss. Adipokines produced by adipose tissue could be one of the mechanisms mediating the association between obesity and periodontal disease. This suggests that obesity may have the potential to modify the host's immunity and inflammatory system.

This project will extend the existing information on the association between obesity and periodontal disease including QoL aspect to a Malaysia population. It will also improve knowledge on the cellular and molecular mechanisms that underpin obesity-periodontal disease relationship. By extension, this study also will cast light on the effects of periodontal interventions for the subgroup population.

DETAILED DESCRIPTION:
Obesity is an epidemic with increasing prevalence in most countries in the Asia Pacific region. It is characterized by abnormal or excessive lipid deposition as a result of chronic disproportion between energy intake and energy outflow. The first Malaysian national estimate in 1996 of obesity was 5.8%. A systematic review reported a marked increase in obesity in 1996, 2003, 2004 and 2006 with 5.5%, 12.2%, 12.3% and 14.0%. Obesity is highest among adults of 40-59 years old, is greater risk in women compared to men and is highest among Indians followed by Malays, Chinese and Aboriginals.

Periodontitis and obesity are both chronic health problems, and an association between the two conditions exists. A positive association was repeatedly demonstrated between obesity and periodontal disease in multiple studies around the world.

Periodontal disease is a chronic oral infection, in which destruction of tooth supporting structures, periodontal ligament and alveolar bone occurs, leading ultimately to tooth loss. Worldwide, the prevalence of periodontitis in the adult population is about 10-15%. In Malaysia, the National Oral Health study reported 90.2% of the adults presented with some forms of periodontal conditions. About 5.5% of these subjects had deep pockets of 6 mm or more.

Periodontal disease, through inflammation and destruction of the periodontium produces a wide range of clinical signs and symptoms, some of which may have a considerable impact on quality of life (QoL). A study conducted using a community sample found a significant association between periodontal disease and quality of life (QoL). They also found that self-reported symptoms of periodontal diseases such as swollen gums, sore gums and receding gums has an apparent impact on the quality of life of the person. With the mechanism of obesity, it is expected that the obese patients may have experienced more severe periodontal diseases and hence they may experience more impact on the quality of life. However, the evidence is still lacking.

Cytokines play a role in the pathogenesis of periodontitis. They play an active role in wound repair and in transient inflammation. They also activate defence mechanisms in which they may give rise to considerable tissue damage in severe inflammation.

Adipose tissue cells namely adipocytes, preadipocytes and macrophages secrete protein signals collectively known as adipokines or adipocytokines. Adipokines are involved in inflammation and the acute-phase response. Production of adipokines increased in obesity, and raised circulating levels of several acute-phase proteins and inflammatory cytokines. This has led to the concept that obese is a state of chronic low-grade systemic inflammation causally link to insulin resistance and metabolic syndrome.

Salivary components comprising of several inflammatory and immune mediators have been identified which are involved in periodontal destruction. Among all the adipokines, resistin which is an adipocyte-derived cytokine is raised in obese mice. In humans, it is suggested that resistin is largely expressed from neutrophils, macrophages, and monocytes other than adipocytes. Resistin is identified as a proinflammatory adipokine that potentially links obesity to diabetes. It is also believed that human resistin stimulates the production and secretion of other proinflammatory molecules like tumor necrosis factor (TNF)-α and interleukin (IL)-12. Studies have shown high levels of resistin in subjects having chronic periodontitis and this may affect systemic health. In a study by Devanoorkar et al., stated that the decrease in the resistin levels was not statistically significant following non-surgical periodontal therapy.

The reason for the interest in GCF/serum levels of resistin in periodontitis lies in the fact that epidemiological research indicates that periodontitis interplays between obesity and diabetes mellitus. It is possible that raised levels of resistin in periodontitis can explain at least in part the link between periodontitis and other chronic inflammatory diseases. Therefore, the overall aim of this systematic review was to provide evidence of resistin biomarker in chronic periodontal disease which might underpin the relationship between periodontal disease, diabetes and obesity. Evidence from case-control studies are all summarized and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Obese i.e. BMI ≥ 30 kg/m2 (WHO 1997)
* Age should be ≥ 30 years old
* Patients should have at least 12 teeth present

Exclusion Criteria:

* Non Malaysian subjects
* Patients who have received periodontal treatment within the past 4 months
* Patients who have been on antibiotics within the past 4 months
* Patients who require prophylactic antibiotic coverage
* Patients who have been on systemic or topical steroidal anti-inflammatory drugs for the past 4 months
* Patients who are pregnant and lactating mothers
* Patients who are mentally handicapped that may interfere with oral hygiene procedures

Min Age: 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2013-02; Primary Completion 2014-01 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
changes in clinical attachment levels (CAL) (mean CAL in mm, as a measure for periodontal parameters) following non surgical periodontal therapy | baseline to 12 weeks

SECONDARY OUTCOMES:
Oral health related quality of life (OHRQoL) | baseline to 12 weeks
salivary resistin (measured in ng/ml) | baseline to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Nor Adinar Baharuddin, DClinDent, Principal Investigator — University of Malaya
Locations (1):
- Faculty of Dentistry, Lembah Pantai, Kuala Lumpur, Malaysia

REFERENCES:
- [Background] Price RA, Reed DR, Guido NJ. Resemblance for body mass index in families of obese African American and European American women. Obes Res. 2000 Aug;8(5):360-6. doi: 10.1038/oby.2000.43. PMID 10968727
- [Background] Asia Pacific Cohort Studies Collaboration. The burden of overweight and obesity in the Asia-Pacific region. Obes Rev. 2007 May;8(3):191-6. doi: 10.1111/j.1467-789X.2006.00292.x. PMID 17444961
- [Background] Khambalia AZ, Seen LS. Trends in overweight and obese adults in Malaysia (1996-2009): a systematic review. Obes Rev. 2010 Jun;11(6):403-12. doi: 10.1111/j.1467-789X.2010.00728.x. Epub 2010 Mar 11. PMID 20233309
- [Background] Kussmann M, Raymond F, Affolter M. OMICS-driven biomarker discovery in nutrition and health. J Biotechnol. 2006 Aug 5;124(4):758-87. doi: 10.1016/j.jbiotec.2006.02.014. Epub 2006 Apr 4. PMID 16600411
- [Background] Suvan J, D'Aiuto F, Moles DR, Petrie A, Donos N. Association between overweight/obesity and periodontitis in adults. A systematic review. Obes Rev. 2011 May;12(5):e381-404. doi: 10.1111/j.1467-789X.2010.00808.x. Epub 2011 Feb 23. PMID 21348914
- [Background] Chaffee BW, Weston SJ. Association between chronic periodontal disease and obesity: a systematic review and meta-analysis. J Periodontol. 2010 Dec;81(12):1708-24. doi: 10.1902/jop.2010.100321. Epub 2010 Aug 19. PMID 20722533
- [Background] Page RC. The role of inflammatory mediators in the pathogenesis of periodontal disease. J Periodontal Res. 1991 May;26(3 Pt 2):230-42. doi: 10.1111/j.1600-0765.1991.tb01649.x. PMID 1679130
- [Background] Yudkin JS, Stehouwer CD, Emeis JJ, Coppack SW. C-reactive protein in healthy subjects: associations with obesity, insulin resistance, and endothelial dysfunction: a potential role for cytokines originating from adipose tissue? Arterioscler Thromb Vasc Biol. 1999 Apr;19(4):972-8. doi: 10.1161/01.atv.19.4.972. PMID 10195925
- [Background] Steppan CM, Bailey ST, Bhat S, Brown EJ, Banerjee RR, Wright CM, Patel HR, Ahima RS, Lazar MA. The hormone resistin links obesity to diabetes. Nature. 2001 Jan 18;409(6818):307-12. doi: 10.1038/35053000. PMID 11201732
- [Background] Hiroshima Y, Bando M, Inagaki Y, Mihara C, Kataoka M, Murata H, Shinohara Y, Nagata T, Kido J. Resistin in gingival crevicular fluid and induction of resistin release by Porphyromonas gingivalis lipopolysaccharide in human neutrophils. J Periodontal Res. 2012 Oct;47(5):554-62. doi: 10.1111/j.1600-0765.2011.01466.x. Epub 2012 Feb 6. PMID 22309231
- [Background] Devanoorkar A, Dwarakanath CD, Gundanavar G, Kathariya R, Patil SR. Evaluation of serum resistin levels in periodontal health and disease and effects of non surgical periodontal therapy on its levels. Dis Markers. 2012;32(5):289-94. doi: 10.1155/2012/153418. PMID 22848926
- [Derived] Basher SS, Saub R, Vaithilingam RD, Safii SH, Daher AM, Al-Bayaty FH, Baharuddin NA. Impact of non-surgical periodontal therapy on OHRQoL in an obese population, a randomised control trial. Health Qual Life Outcomes. 2017 Nov 21;15(1):225. doi: 10.1186/s12955-017-0793-7. PMID 29157276